CLINICAL TRIAL: NCT01190930
Title: Treatment of Patients With Newly Diagnosed Standard Risk B-Lymphoblastic Leukemia (B-ALL) or Localized B-Lineage Lymphoblastic Lymphoma (B-LLy)
Brief Title: Risk-Adapted Chemotherapy in Treating Younger Patients With Newly Diagnosed Standard-Risk Acute Lymphoblastic Leukemia or Localized B-Lineage Lymphoblastic Lymphoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AALL0932; NCI-2011-02599 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000683227; 11-00080; AALL0932 (Other: Children's Oncology Group); AALL0932 (Other: CTEP); U10CA180886 (NIH); U10CA098543 (NIH)
Record Dates: First submitted 2010-08-27; First posted 2010-08-30 (Estimated); Results first posted 2020-06-23 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Acute Lymphoblastic Leukemia; Adult B Lymphoblastic Lymphoma; Ann Arbor Stage I B Lymphoblastic Lymphoma; Ann Arbor Stage II B Lymphoblastic Lymphoma; Childhood B Acute Lymphoblastic Leukemia; Childhood B Acute Lymphoblastic Leukemia With t(9;22)(q34.1;q11.2); BCR-ABL1; Childhood B Lymphoblastic Lymphoma; Down Syndrome; Hypodiploid B Acute Lymphoblastic Leukemia; Philadelphia Chromosome Positive
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor B-Cell Lymphoblastic Leukemia-Lymphoma; Down Syndrome | interventions — Cyclophosphamide; Cytarabine; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Doxorubicin; Leucovorin; Mercaptopurine; azathiopurine; Methotrexate; merphos; pegaspargase; Thioguanine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Arm A (risk-adapted chemotherapy) (Experimental): Patients receive vincristine sulfate IV on days 1, 29, and 57; dexamethasone PO BID on days 1-5, 29-33, and 57-61; methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78; mercaptopurine PO on days 1-84; and IT methotrexate on day 1.
  Interventions: Drug: Dexamethasone; Other: Laboratory Biomarker Analysis; Drug: Mercaptopurine; Drug: Methotrexate; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Vincristine Sulfate
- Arm B (risk-adapted chemotherapy) (Experimental): Patients receive vincristine sulfate IV on days 1, 29, and 57; dexamethasone PO BID on days 1-5, 29-33, and 57-61; higher-dose methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78; mercaptopurine PO on days 1-84; and IT methotrexate on day 1.
  Interventions: Drug: Dexamethasone; Other: Laboratory Biomarker Analysis; Drug: Mercaptopurine; Drug: Methotrexate; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Vincristine Sulfate
- Arm B-LLy (4-week cycle maintenance) (Experimental): See Detailed Description.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Thioguanine; Drug: Vincristine Sulfate
- Arm C (risk-adapted chemotherapy) (Experimental): Patients receive vincristine sulfate IV on day 1; dexamethasone PO BID on days 1-5; methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78; mercaptopurine PO on days 1-84; and IT methotrexate on day 1.
  Interventions: Drug: Dexamethasone; Other: Laboratory Biomarker Analysis; Drug: Mercaptopurine; Drug: Methotrexate; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Vincristine Sulfate
- Arm D (risk-adapted chemotherapy) (Experimental): Patients receive vincristine sulfate IV on day 1; dexamethasone PO BID on days 1-5; higher-dose methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78; mercaptopurine PO on days 1-84; and IT methotrexate on day 1.
  Interventions: Drug: Dexamethasone; Other: Laboratory Biomarker Analysis; Drug: Mercaptopurine; Drug: Methotrexate; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Vincristine Sulfate
- Arm LR-C (risk-adapted chemotherapy) (Experimental): Patients receive consolidation, interim maintenance I, delayed intensification, interim maintenance II, and maintenance therapy. See detailed description.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Thioguanine; Drug: Vincristine Sulfate
- Arm LR-M (risk-adapted chemotherapy) (Experimental): Patients receive consolidation and maintenance therapy. See detailed description.
  Interventions: Drug: Dexamethasone; Other: Laboratory Biomarker Analysis; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Methotrexate; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Vincristine Sulfate
- Arm SR DS (12-week cycle maintenance) (Experimental): See Detailed Description
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Thioguanine; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
  Arms: Arm B-LLy (4-week cycle maintenance); Arm LR-C (risk-adapted chemotherapy); Arm SR DS (12-week cycle maintenance)
Drug: Cytarabine — Given IT, IV, or SC
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
  Arms: Arm B-LLy (4-week cycle maintenance); Arm LR-C (risk-adapted chemotherapy); Arm SR DS (12-week cycle maintenance)
Drug: Dexamethasone — Given orally (PO) or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; LenaDex; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
  Arms: Arm B-LLy (4-week cycle maintenance); Arm LR-C (risk-adapted chemotherapy); Arm SR DS (12-week cycle maintenance)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Leucovorin Calcium — Given PO
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
  Arms: Arm B-LLy (4-week cycle maintenance); Arm LR-M (risk-adapted chemotherapy); Arm SR DS (12-week cycle maintenance)
Drug: Mercaptopurine — Given PO
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; Bw 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
Drug: Methotrexate — Given IT, PO, or IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Jylamvo; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Pegaspargase — Given IV
  Other Names: L-Asparaginase with Polyethylene Glycol; Oncaspar; Oncaspar-IV; PEG-Asparaginase; PEG-L-Asparaginase; PEG-L-Asparaginase (Enzon - Kyowa Hakko); PEGLA; Polyethylene Glycol L-Asparaginase; Polyethylene Glycol-L-Asparaginase
  Arms: Arm B-LLy (4-week cycle maintenance); Arm LR-C (risk-adapted chemotherapy); Arm SR DS (12-week cycle maintenance)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Thioguanine — Given PO
  Other Names: 2-Amino 6MP; 2-Amino-1,7-dihydro-6H-purine-6-thione; 2-Amino-6-mercaptopurine; 2-Amino-6-purinethiol; 2-Aminopurin-6-thiol; 2-Aminopurine-6(1H)-thione; 2-Aminopurine-6-thiol; 2-Aminopurine-6-thiol Hemihydrate; 2-Mercapto-6-aminopurine; 6-Amino-2-mercaptopurine; 6-Mercapto-2-aminopurine; 6-Mercaptoguanine; 6-TG; 6H-Purine-6-thione, 2-amino-1,7-dihydro- (9CI); BW 5071; Lanvis; Tabloid; Thioguanine Hemihydrate; Thioguanine Hydrate; Tioguanin; Tioguanine; Wellcome U3B; WR-1141; X 27
  Arms: Arm B-LLy (4-week cycle maintenance); Arm LR-C (risk-adapted chemotherapy); Arm SR DS (12-week cycle maintenance)
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This partially randomized phase III trial studies the side effects of different combinations of risk-adapted chemotherapy regimens and how well they work in treating younger patients with newly diagnosed standard-risk acute lymphoblastic leukemia or B-lineage lymphoblastic lymphoma that is found only in the tissue or organ where it began (localized). Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving more than one drug (combination chemotherapy), giving the drugs in different doses, and giving the drugs in different combinations may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

l. To determine if a maintenance regimen containing weekly oral methotrexate at 40 mg/m^2/week will result in an improved disease free survival (DFS) compared to that containing weekly oral methotrexate at 20 mg/m^2/week in the average-risk (AR) subset of patients with standard-risk B-precursor acute lymphoblastic leukemia (ALL). (Complete effective January 13, 2017) II. To determine whether a reduced-pulses maintenance regimen with vincristine (vincristine sulfate)/dexamethasone pulses delivered every 12 weeks can be used without adversely impacting DFS as compared to pulses given every 4 weeks in the AR subset of patients with standard risk B-precursor ALL.

III. To confirm that patients in the low-risk (LR) subset of standard risk B-precursor ALL, based on clinical and cytogenetic features and minimal residual disease (MRD) criteria, can attain a 5 year DFS of at least 95% with either a P9904 based regimen that includes 6 courses of intermediate dose (1 g/m^2 over 24 hours) methotrexate without alkylating agents or anthracyclines (Arm LR-M), or an outpatient based regimen identical to that of AR patients with reduced vincristine/dexamethasone pulses at 12 week intervals during maintenance (Arm LR-C).

IV. To provide standardized treatment and enhanced supportive care to children with standard-risk (SR) Down syndrome B-ALL in order to improve outcomes and facilitate further study of this biologically and clinically unique patient subgroup.

V. To improve understanding of the biology of localized B-lineage lymphoblastic lymphoma (B-LLy) and Down syndrome (DS) B-LLy by obtaining biologic data, including fluorescence in situ hybridization (FISH) for recurrent cytogenetic lesions on paraffin specimen, and banking tissue for future research.

VI. To describe the 5-year event free survival (EFS) and overall survival (OS) of patients with Murphy stage I and II B-LLy receiving modified AR B-ALL therapy.

SECONDARY OBJECTIVES:

I. To assess the burden of AR B-ALL therapy as measured by surveys of the child's quality of life, missed days of school/daycare/work by children and parents, family functioning, parental perception of the child's health vulnerability, physical functioning, and emotional distress, 1) overall at different time points during and at the end of therapy, and by 2) comparing children randomized to every 4 week vs. every 12 week dexamethasone/vincristine pulses during maintenance. (Closed to accrual as of April 19, 2013) II. To characterize the onset, severity, and natural history of vincristine associated neuropathy by physical therapists (or occupational therapists) in children undergoing therapy for AR B-ALL, 1) overall at different time points during and at the end of therapy, and by 2) comparing children randomized to every 4 week vs. every 12 week dexamethasone/vincristine pulses during maintenance. (Closed to accrual as of March 15, 2013)

TERTIARY OBJECTIVES:

I. To explore the correlation of minimal marrow disease (MMD) at diagnosis and outcome for patients with B-LLy. (Closed effective Amendment #5)

OUTLINE:

All patients receive induction therapy comprising intrathecal (IT) cytarabine on day 1; vincristine sulfate IV on days 1, 8, 15, and 22; dexamethasone orally (PO) or IV twice daily (BID) on days 1-28; pegaspargase IV over 1-2 hours on day 4; and IT methotrexate* on days 8 and 29. Patients with Philadelphia chromosome-positive disease are eligible to transfer to COG-AALL0622 by day 15 of induction therapy and patients with high-risk (HR) or very high-risk (VHR) disease are eligible to transfer to a COG HR or VHR trial at the end of induction therapy. Patients with standard-risk disease with Down syndrome (DS) who have bone marrow minimal residual disease 0.01% are eligible to transfer to the DS stratum of the HR trial. Patients with induction failure (defined as M3 [> 25% lymphoblasts] on day 29) may be eligible for the COG VHR-acute lymphoblastic leukemia study.

NOTE: *Patients with DS also receive oral leucovorin calcium every 12 hours on days 10-11 and 31-32.

STANDARD-RISK WITH DOWN SYNDROME:

Consolidation therapy (4 weeks): Patients receive vincristine sulfate IV on day 1; mercaptopurine PO on days 1-28; IT methotrexate on days 1, 8, and 15; and leucovorin calcium PO every 12 hours on days 3-4, 10-11, and 17-18. Interim maintenance I therapy (8 weeks): Patients receive vincristine sulfate IV and methotrexate IV over 2-15 minutes on days 1, 11, 21, 31, and 41; IT methotrexate on day 31; and leucovorin calcium PO every 12 hours on days 36-34. Delayed-intensification therapy (8 weeks): Patients receive dexamethasone PO or IV BID on days 1-7 and 15-21; vincristine sulfate IV and doxorubicin hydrochloride IV over 1-15 minutes on days 1, 8, and 15; pegaspargase IV over 1-2 hours on day 4; cyclophosphamide IV over 30-60 minutes on day 29; thioguanine PO on days 29-42; cytarabine IV over 1-30 minutes or subcutaneously (SC) on days 29-32 and 33-39; IT methotrexate on days 1 and 29; and leucovorin calcium PO every 12 hours on days 3-4 and 31-32. Interim maintenance II therapy (8 weeks): Patients receive vincristine sulfate IV and methotrexate IV over 2-15 minutes on days 1, 11, 21, 31, and 41; IT methotrexate on days 1 and 31; and leucovorin calcium PO every 12 hours on days 3-4 and 33-34. Maintenance therapy: Patients receive vincristine sulfate IV on day 1; dexamethasone PO BID on days 1-5; methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78; mercaptopurine PO on days 1-84; and IT methotrexate on day 1. Courses repeat every 12 weeks for 2 years (timed from the start of interim maintenance I therapy).

B-LLy:

Consolidation therapy (4 weeks): Patients receive vincristine sulfate IV on day 1; mercaptopurine PO on days 1-28; IT methotrexate on days 1, 8, and 15; and leucovorin calcium PO every 12 hours on days 3-4, 10-11, and 17-18. Interim maintenance I therapy (8 weeks): Patients receive vincristine sulfate IV and methotrexate IV over 2-15 minutes on days 1, 11, 21, 31, and 41; IT methotrexate on day 31; and leucovorin calcium PO every 12 hours on days 36-34. Delayed-intensification therapy (8 weeks): Patients receive dexamethasone PO or IV BID on days 1-7 and 15-21; vincristine sulfate IV and doxorubicin hydrochloride IV over 1-15 minutes on days 1, 8, and 15; pegaspargase IV over 1-2 hours on day 4; cyclophosphamide IV over 30-60 minutes on day 29; thioguanine PO on days 29-42; cytarabine IV over 1-30 minutes or subcutaneously (SC) on days 29-32 and 33-39; IT methotrexate on days 1 and 29; and leucovorin calcium PO every 12 hours on days 3-4 and 31-32. Interim maintenance II therapy (8 weeks): Patients receive vincristine sulfate IV and methotrexate IV over 2-15 minutes on days 1, 11, 21, 31, and 41; IT methotrexate on days 1 and 31; and leucovorin calcium PO every 12 hours on days 3-4 and 33-34. Maintenance therapy: Patients receive vincristine sulfate IV on day 1; dexamethasone PO BID on days 1-5; methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78; mercaptopurine PO on days 1-84; and IT methotrexate on day 1. Courses repeat every 4 weeks for 2 years (timed from the start of interim maintenance I therapy).

AVERAGE-RISK:

Consolidation therapy (4 weeks): Patients receive vincristine sulfate IV on day 1; mercaptopurine PO on days 1-28; and IT methotrexate on days 1, 8, and 15.Interim maintenance I therapy (8 weeks): Patients receive vincristine sulfate IV and methotrexate IV over 2-15 minutes on days 1, 11, 21, 31, and 41 and IT methotrexate on day 31. Delayed intensification therapy (8 weeks): Patients receive dexamethasone PO or IV BID on days 1-7 and 15-21; vincristine sulfate IV and doxorubicin hydrochloride IV over 1-15 minutes on days 1, 8, and 15; pegaspargase IV over 1-2 hours on day 4; cyclophosphamide IV over 30-60 minutes on day 29; thioguanine PO on days 29-42; cytarabine IV over 1-30 minutes or SC on days 29-32 and 36-39; and IT methotrexate on days 1 and 29. Interim maintenance II therapy (8 weeks): Patients receive vincristine sulfate IV and methotrexate IV over 2-15 minutes on days 1, 11, 21, 31, and 41 and IT methotrexate on days 1 and 31. Maintenance therapy: Patients are randomized to 1 of 4 maintenance therapy treatment arms.

Arm A: Patients receive vincristine sulfate IV on days 1, 29, and 57; dexamethasone PO BID on days 1-5, 29-33, and 57-61; methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78; mercaptopurine PO on days 1-84; and IT methotrexate on day 1.

Arm B: Patients receive vincristine sulfate IV on days 1, 29, and 57; dexamethasone PO BID on days 1-5, 29-33, and 57-61; higher-dose methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78; mercaptopurine PO on days 1-84; and IT methotrexate on day 1.

Arm C: Patients receive vincristine sulfate IV on day 1; dexamethasone PO BID on days 1-5; methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78; mercaptopurine PO on days 1-84; and IT methotrexate on day 1.

Arm D: Patients receive vincristine sulfate IV on day 1; dexamethasone PO BID on days 1-5; higher-dose methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78; mercaptopurine PO on days 1-84; and IT methotrexate on day 1.

In all arms, maintenance therapy courses repeat every 12 weeks for 2 years for girls and for 3 years for boys (timed from the start of interim maintenance I therapy).

LOW-RISK: Patients are randomized to 1 of 2 treatment arms.

Arm I (LR-M): Consolidation therapy (19 weeks): Beginning one week after completion of induction therapy, patients receive vincristine sulfate IV on days 15, 22, 78, and 85; methotrexate IV over 24 hours and IT methotrexate on days 8, 29, 50, 71, 92, and 113; leucovorin calcium PO or IV on days 9-10, 30-31, 51-52, 72-73, 93-94, and 114-115; dexamethasone PO BID or IV on days 15-21 and 78-84; and PO mercaptopurine on days 1-133.Maintenance therapy: Patients receive vincristine sulfate IV on days 1 and 8; dexamethasone PO BID on days 1-7; methotrexate* PO on days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, 85, 92, 99, and 106; and mercaptopurine PO on days 1-112. Courses repeat every 16 weeks. Patients also receive IT methotrexate on days 1 and 85 (courses 1 and 4), day 57 (courses 2 and 5), or day 29 (courses 3 and 6). Patients then receive course 7 comprising vincristine sulfate IV on days 1 and 8; dexamethasone PO BID on days 1-7; methotrexate PO on days 1, 8, 15, 22, 29, 36, 43, 50, 57, and 64; and mercaptopurine PO on days 1-70. Treatment continues for 2 and Â½ years (timed from the date of diagnosis).NOTE: *Patients do not receive methotrexate PO on the days that they receive IT methotrexate.

Arm II (LR-C): Consolidation therapy (4 weeks): Patients receive vincristine sulfate IV on day 1; oral mercaptopurine on days 1-28; and IT methotrexate on days 1, 8, and 15. Interim maintenance I therapy (8 weeks): Patients receive vincristine sulfate IV and methotrexate IV over 2-15 minutes on days 1, 11, 21, 31, and 41 and IT methotrexate on day 31. Delayed-intensification therapy (8 weeks): Patients receive dexamethasone PO or IV BID on days 1-7 and 15-21; vincristine sulfate IV and doxorubicin hydrochloride IV over 1-15 minutes on days 1, 8, and 15; pegaspargase IV over 1-2 hours on day 4; cyclophosphamide IV over 30-60 minutes on day 29; thioguanine PO on days 29-42; cytarabine IV over 1-30 minutes or SC on days 29-32 and 36-39; and IT methotrexate on days 1 and 29.Interim maintenance II therapy (8 weeks): Patients receive vincristine sulfate IV and methotrexate IV over 2-15 minutes on days 1, 11, 21, 31, and 41 and IT methotrexate on days 1 and 31. Maintenance therapy: Patients receive vincristine sulfate IV on day 1; dexamethasone PO BID on days 1-5; methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78; mercaptopurine PO on days 1-84; and IT methotrexate on day 1. Courses repeat every 12 weeks for 2 years for girls and for 3 years for boys (timed from the start of interim maintenance I therapy).

After completion of study treatment, patients are followed up periodically for 10 years from study entry.

ELIGIBILITY:
Inclusion Criteria:

* B-ALL patients must be enrolled on AALL08B1 or APEC14B1 (if open for the classification of newly diagnosed ALL patients) prior to treatment and enrollment on AALL0932

  * Note: B-LLy patients are not eligible for AALL08B1, and can enroll directly onto AALL0932
* B-ALL patients must have an initial white blood cell count < 50,000/uL
* Patients must have newly diagnosed National Cancer Institute (NCI) Standard Risk B-ALL or B-LLy Murphy stages I or II; patients with Down syndrome are also eligible

  * Note: for B-LLy patients with tissue available for flow cytometry, the criterion for diagnosis should be analogous to B-ALL; for tissue processed by other means (i.e. paraffin blocks), the methodology and criteria for immunophenotypic analysis to establish the diagnosis of B-LLy defined by the submitting institution will be accepted
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and NCI requirements for human studies must be met

Exclusion Criteria:

* With the exception of steroid pretreatment (defined below) or the administration of intrathecal cytarabine, patients must not have received any prior cytotoxic chemotherapy for either the current diagnosis of B-ALL or B-LLy or for any cancer diagnosed prior to initiation of protocol therapy on AALL0932

  * Patients receiving prior steroid therapy may be eligible for AALL0932
* Patients with central nervous system 3 (CNS3) leukemia

  * CNS status must be known prior to enrollment; (Note: the CNS status must be determined based on a sample obtained prior to administration of any systemic or intrathecal chemotherapy, except for steroid pretreatment); B-LLy patients with CNS3 disease are not eligible for this protocol or the COG HR ALL protocol; it is recommended that intrathecal cytarabine be administered at the time of the diagnostic lumbar puncture; this is usually done at the time of the diagnostic bone marrow or venous line placement to avoid a second lumbar puncture; this is allowed prior to registration; systemic chemotherapy must begin within 72 hours of the first dose of intrathecal therapy
* B-ALL patients with testicular leukemia are not eligible for AALL0932
* For B-LLy patients the following additional exclusion criteria apply:

  * T-lymphoblastic lymphoma
  * Morphologically unclassifiable lymphoma
  * Absence of both B-cell and T-cell phenotype markers in a case submitted as lymphoblastic lymphoma
  * CNS3-positive disease or testicular involvement
  * M2 (5% - 25% blasts) or M3 (> 25% blasts) marrow
  * Female patients who are pregnant are ineligible
  * Lactating females are not eligible unless they have agreed not to breastfeed their infants
  * Female patients of childbearing potential are not eligible unless a negative pregnancy test result has been obtained
  * Sexually active patients of reproductive potential are not eligible unless they have agreed to use an effective contraceptive method for the duration of their study participation

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9350 (Actual)
Dates: Start 2010-08-09 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2028-03-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Anne L Angiolillo, Principal Investigator — Children's Oncology Group
Locations (243):
- United States (213):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Vannie Cook Children's Clinic, McAllen, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (9):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Children's Hospital-Brisbane, Herston, Queensland
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Monash Medical Center-Clayton Campus, Clayton, Victoria
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (14):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Our Lady's Children's Hospital, Dublin, Co Dublin, Ireland
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- Puerto Rico (2):
  - San Jorge Children's Hospital, San Juan
  - University Pediatric Hospital, San Juan
- Switzerland (2):
  - Swiss Pediatric Oncology Group - Geneva, Geneva
  - Swiss Pediatric Oncology Group - Lausanne, Lausanne

IPD SHARING:
Plan to Share IPD: Yes
Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive

REFERENCES:
- [Derived] Chen W, Chang TC, Rabin KR, Raetz EA, Devidas M, Hunger SP, Ramirez NC, Mullighan CG, Loh ML, Wu G. Performance of Two-Phase Designs for the Time-to-Event Outcome and a Case Study Assessing the Relapse Risk Associated With B-ALL Subtypes. JCO Clin Cancer Inform. 2025 May;9:e2400223. doi: 10.1200/CCI-24-00223. Epub 2025 May 2. PMID 40315406
- [Derived] Chang TC, Chen W, Qu C, Cheng Z, Hedges D, Elsayed A, Pounds SB, Shago M, Rabin KR, Raetz EA, Devidas M, Cheng C, Angiolillo A, Baviskar P, Borowitz M, Burke MJ, Carroll A, Carroll WL, Chen IM, Harvey R, Heerema N, Iacobucci I, Wang JR, Jeha S, Larsen E, Mattano L, Maloney K, Pui CH, Ramirez NC, Salzer W, Willman C, Winick N, Wood B, Hunger SP, Wu G, Mullighan CG, Loh ML. Genomic Determinants of Outcome in Acute Lymphoblastic Leukemia. J Clin Oncol. 2024 Oct 10;42(29):3491-3503. doi: 10.1200/JCO.23.02238. Epub 2024 Aug 9. PMID 39121442
- [Derived] Rabin KR, Devidas M, Chen Z, Ji L, Kairalla J, Hitzler JK, Yang JJ, Carroll AJ, Heerema NA, Borowitz MJ, Wood BL, Roberts KG, Mullighan CG, Harvey RC, Chen IM, Willman CL, Reshmi SC, Gastier-Foster JM, Bhojwani D, Rheingold SR, Maloney KW, Mattano LA, Larsen EC, Schore RJ, Burke MJ, Salzer WL, Winick NJ, Carroll WL, Raetz EA, Loh ML, Hunger SP, Angiolillo AL. Outcomes in Children, Adolescents, and Young Adults With Down Syndrome and ALL: A Report From the Children's Oncology Group. J Clin Oncol. 2024 Jan 10;42(2):218-227. doi: 10.1200/JCO.23.00389. Epub 2023 Oct 27. PMID 37890117
- [Derived] Angiolillo AL, Schore RJ, Kairalla JA, Devidas M, Rabin KR, Zweidler-McKay P, Borowitz MJ, Wood B, Carroll AJ, Heerema NA, Relling MV, Hitzler J, Lane AR, Maloney KW, Wang C, Bassal M, Carroll WL, Winick NJ, Raetz EA, Loh ML, Hunger SP. Excellent Outcomes With Reduced Frequency of Vincristine and Dexamethasone Pulses in Standard-Risk B-Lymphoblastic Leukemia: Results From Children's Oncology Group AALL0932. J Clin Oncol. 2021 May 1;39(13):1437-1447. doi: 10.1200/JCO.20.00494. Epub 2021 Jan 7. PMID 33411585
- Available data/document: Individual Participant Data Set — https://nctn-data-archive.nci.nih.gov/ — Available IPD/Information: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Newly Diagnosed Standard Risk B-Lymphoblastic Leukemia (B-ALL) or Localized B-lineage Lymphoblastic Lymphoma (B-LLy)
Pre-assignment Details: Patients were stratified between 2 disease groups (B-ALL and B-LLY) for Induction and then risk assigned treatment based upon the patient's response.
Groups:
- B-ALL: All patients receive induction therapy comprising intrathecal (IT) cytarabine on day 1; vincristine sulfate IV on days 1, 8, 15, and 22; dexamethasone orally (PO) or IV twice daily (BID) on days 1-28; pegaspargase IV over 1-2 hours on day 4; and IT methotrexate on days 8 and 29. Patients with DS also receive leucovorin calcium every 12 hours on days 10-11 and 21-32. Patients with Philadelphia chromosome-positive disease are eligible to transfer to COG-AALL0622 by day 15 of induction therapy and patients with high-risk (HR) or very high-risk (VHR) disease are eligible to transfer to a COG HR or VHR trial at the end of induction therapy. Patients with standard-risk disease with Down syndrome (DS) who have bone marrow minimal residual disease 0.01% are eligible to transfer to the DS stratum of the HR trial. Patients with induction failure (defined as M3 [> 25% lymphoblasts] on day 29) may be eligible for the COG VHR-acute lymphoblastic leukemia study.
- B-LLy: Induction: same trt as B-ALL; Consolidation (4 wks): vincristine sulfate day 1; mercaptopurine days 1-28; IT methotrexate (MTX) days 1/8/15; leucovorin calcium days 3-4,10-11,17-18 Interim maintenance I (8 wks): vincristine sulfate and MTX 2-15 min days 1/11/21/31/41; IT MTX day 31; leucovorin calcium days 33-34 Delayed-intensification (8 wks): dexamethasone days 1-7 and 15-21; vincristine sulfate and doxorubicin hydrochloride on days 1/8/15; pegaspargase 1-2 hrs day 4; cyclophosphamide day 29; thioguanine days 29-42; cytarabine 29-32, 33-39; IT MTX days 1/29; and leucovorin calcium days 3-4, 31-32 Interim maintenance II (8 wks): vincristine sulfate and MTX days 1/11/21/31/41; IT MTX days 1/31; and leucovorin calcium days 3-4, 33/34 Maintenance: vincristine sulfate day 1; dexamethasone days 1-5; MTX weekly days 8-78; mercaptopurine days 1-84; and IT MTX day 1. Courses repeat every 4 wks for 2 yrs (from the start of IMI therapy).
- B-ALL Average Risk: Consolidation (4 wks): vincristine (VIN) day (d) 1; mercaptopurine (MP) d 1-28; IT MTX d 1/8/15; leucovorin (LV) d 3-4/10-11/17-18 Int. maint. I (8 wks): VIN and MTX d 1/11/21/31/41; IT MTX d 31; LV d 33-34 Delayed-intensification (8 wks): dexamethasone (DEX) d 1-7/15-21; VIN and doxorubicin d 1/8/15; pegaspargase d 4; cyclophosphamide d 29; thioguanine d 29-42; cytarabine d 29-32/33-39; IT MTX d 1/29; LV d 3-4/31-32 Int. maint. II (8 wks): VIN and MTX d 1/11/21/31/41; IT MTX d 1/31; LV d 3-4/33-34
- Standard Risk With Down Syndrome: Consolidation (4 w): vincristine (VIN) d1; MP d1-28; IT methotrexate (MTX) d1/8/15; leucovorin (LV) d3-4/10-11/17-18 Interim maintenance I (8 wks): VIN & IV MTX d1/11/21/31/41; IT MTX d31; LV d36-34 Delayed-intensification (8 wks): Patients receive dexamethasone (DEX) d1-7/15-21; VIN & doxorubicin d1/8/15; pegaspargase d4; cyclophosphamide d29; thioguanine d 29-42; cytarabine d29-32/33-39; IT MTX d1/29; and LV d3-4/31-32 Interim maintenance II (8 wks): VIN & IV MTX d1/11/21/31/41; IT MTX d1/31; and LV d3-4/33-34 Maintenance: VIN d1; DEX d1-5; PO MTX wkly d8-78; MP d1-84; and IT MTX d1. Courses repeat every 12 wks for 2 years (timed from the start of interim maintenance I therapy).
- B-ALL Low Risk Arm I (LR-M): Consolidation (19 w): vincristine (VIN) day(d) 15/22/78/85; IV/IT methotrexate (MTX) d8/29/50/71/92/113; leucovorin (LV) d9-10/30-31/51-52/72-73/93-94/114-115; dexamethasone (DEX) d15-21/78-84; mercaptopurine (MP) d 1-133. Maint.: VIN d1/8; DEX d1-7; MTX* PO wkly d1-106; MP d 1-112. Repeat every 16 w until 2.5 yrs from dx. IT MTX d1/85 (course 1&4), d 57 (course 2&5), d29 (course 3&6). Course 7: VIN d1/8; DEX d 1-7; MTX PO wkly d8-64; and MP d1-70. *Patients do not receive MTX PO on d w/ IT MTX.
- B-ALL Low Risk Arm II (LR-C): Consolidation (4 w): VIN d1; MP d1-28; IT MTX d1/8/15 Interim Maint. I (8 w): VIN & IV MTX d1/11/21/31/41; IT MTX d31 Delayed-intensification (8 w): DEX d1-7/15-21; VIN & doxorubicin d1/8/15; pegaspargase d4; cyclophosphamide d29; thioguanine d 29-42; cytarabine d29-32/36-39; IT MTX d1/29 Interim Maint. II (8 w): VIN & IV MTX d1/11/21/31/41; IT MTX d1/31 Maint.: VIN d1; DEX d1-5; MTX PO wkly d22-78; MP d 1-84; IT MTX d1. Rpt every 12 w for 2 yrs:girls, 3 yrs:boys from start IM1
- B-ALL Average Risk-Arm A: Maintenance: repeat every 12 wks for 2 yrs (girls), 3 yrs (boys) from start IM1: VIN d 1/29/57; DEX d 1-5/29-33/57-61; MTX weekly d 8-78; MP d 1+P8:W8-84; and IT MTX d 1
- B-ALL Average Risk-Arm B: Maintenance: repeat every 12 wks for 2 yrs (girls), 3 yrs (boys) from start IM1: VIN d 1/29/57; DEX d 1-5/29-33/57-61; high-dose (HD) MTX weekly d 8-78; MP d 1-84; and IT MTX d 1
- B-ALL Average Risk-Arm C: Maintenance: repeat every 12 wks for 2 yrs (girls), 3 yrs (boys) from start IM1: VIN d 1; DEX d 1-5; MTX weekly d 8-78; MP d 1-84; IT MTX d 1
- B-ALL Average Risk-Arm D: Maintenance: repeat every 12 wks for 2 yrs (girls), 3 yrs (boys) from start IM1: VIN d 1; DEX d 1-5; HD MTX weekly d 8-78; MP d 1-84; IT MTX d 1
Period: Induction
Arm/Group | B-ALL | B-LLy | B-ALL Average Risk | Standard Risk With Down Syndrome | B-ALL Low Risk Arm I (LR-M) | B-ALL Low Risk Arm II (LR-C) | B-ALL Average Risk-Arm A | B-ALL Average Risk-Arm B | B-ALL Average Risk-Arm C | B-ALL Average Risk-Arm D
Started | 9298 | 52 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3949 | 43 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 5349 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 17 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 34 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 125 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Refusal | 235 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Inevaluable | 23 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — BM MRD >= 0.01% on Day 29 of Induction | 61 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — High Risk Downs | 80 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Enrollment onto another COG Protocol | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Average Risk | 1847 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — High Risk | 1227 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Low Risk | 443 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Very High Risk | 1012 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Philadelphia chromosome-positive | 99 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Incomplete Induction data | 63 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — No treatment | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Ineligible | 69 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Post Induction Pre-Maintenance
Arm/Group | B-ALL | B-LLy | B-ALL Average Risk | Standard Risk With Down Syndrome | B-ALL Low Risk Arm I (LR-M) | B-ALL Low Risk Arm II (LR-C) | B-ALL Average Risk-Arm A | B-ALL Average Risk-Arm B | B-ALL Average Risk-Arm C | B-ALL Average Risk-Arm D
Started | 0 | 43 | 3122 | 224 | 301 | 302 | 0 | 0 | 0 | 0
Completed | 0 | 37 | 2364 | 207 | 296 | 296 | 0 | 0 | 0 | 0
Not Completed | 0 | 6 | 758 | 17 | 5 | 6 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 8 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 35 | 7 | 5 | 3 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 5 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Refusal | 0 | 2 | 694 | 4 | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Inevaluable | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — CR failure at the end of consolidation | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Relapse | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Maintenance
Arm/Group | B-ALL | B-LLy | B-ALL Average Risk | Standard Risk With Down Syndrome | B-ALL Low Risk Arm I (LR-M) | B-ALL Low Risk Arm II (LR-C) | B-ALL Average Risk-Arm A | B-ALL Average Risk-Arm B | B-ALL Average Risk-Arm C | B-ALL Average Risk-Arm D
Started | 0 | 37 | 0 | 207 | 296 | 296 | 600 | 586 | 586 | 592
Completed | 0 | 27 | 0 | 167 | 287 | 284 | 574 | 540 | 540 | 555
Not Completed | 0 | 10 | 0 | 40 | 9 | 12 | 26 | 46 | 46 | 37
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 3 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 5 | 9 | 4 | 8 | 8 | 10 | 17
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 4 | 1
Not completed — Refusal | 0 | 1 | 0 | 2 | 0 | 4 | 5 | 17 | 13 | 6
Not completed — second malignant neoplasm | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Inevaluable | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Not completed — Enrollment onto another COG Protocol | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Relapse | 0 | 0 | 0 | 2 | 0 | 1 | 6 | 13 | 11 | 11
Not completed — Still on therapy | 0 | 8 | 0 | 29 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data were collected according to the Arms from the Induction period (1. B-ALL; 2. B-LLy)
Groups:
- B-ALL: All B-ALL patients
- B-LLy: All B-LLy patients
- Total: Total of all reporting groups
Arm/Group | B-ALL | B-LLy | Total
Number analyzed (Participants) | 9298 | 52 | 9350
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9298 | 51 | 9349
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.57 (2.12) | 9.19 (4.40) | 4.59 (2.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4294 | 27 | 4321
  Male | 5004 | 25 | 5029
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2132 | 15 | 2147
  Not Hispanic or Latino | 6726 | 35 | 6761
  Unknown or Not Reported | 440 | 2 | 442
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 94 | 0 | 94
  Asian | 430 | 1 | 431
  Native Hawaiian or Other Pacific Islander | 48 | 0 | 48
  Black or African American | 501 | 1 | 502
  White | 6857 | 40 | 6897
  More than one race | 60 | 1 | 61
  Unknown or Not Reported | 1308 | 9 | 1317

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival (DFS) in Average Risk (AR) Patients Based on the Methotrexate Dose Randomization
Description: DFS is calculated as the time from randomization at the end of interim maintenance II to first event (relapse, second malignancy, remission death) or date of last contact. Five year DFS estimates will be calculated from the point of randomization for both groups. Two-sided 95% confidence intervals will be calculated.
Time Frame: 5.7 years
Population: Average Risk (AR) B-ALL patients who were randomized and started maintenance
Measure: Number (95% Confidence Interval); unit: percent probability
Groups:
- B-ALL Average Risk: MTX 20 mg/m^2/Week Starting Dose; B-ALL Average Risk: MTX 40 mg/m^2/Week Starting Dose: Cons. (4 wks): vincristine (VIN) day (d) 1; mercaptopurine (MP) d 1-28; IT MTX d 1/8/15; leucovorin (LV) d 3-4/10-11/17-18 Int. maint. I (8 wks): VIN and MTX d 1/11/21/31/41; IT MTX d 31; LV d 33-34 Delayed-intensification (8 wks): dexamethasone (DEX) d 1-7/15-21; VIN and doxorubicin d 1/8/15; pegaspargase d 4; cyclophosphamide d 29; thioguanine d 29-42; cytarabine d 29-32/33-39; IT MTX d 1/29; LV d 3-4/31-32 Int. maint. II (8 wks): VIN and MTX d 1/11/21/31/41; IT MTX d 1/31; LV d 3-4/33-34 Maintenance: repeat every 12 wks for 2 yrs (girls), 3 yrs (boys) from start IM1 Arm A: VIN d 1/29/57; DEX d 1-5/29-33/57-61; MTX weekly d 8-78; MP d 1-84; and IT MTX d 1 Arm B: VIN d 1/29/57; DEX d 1-5/29-33/57-61; high-dose (HD) MTX weekly d 8-78; MP d 1-84; and IT MTX d 1 Arm C: VIN d 1; DEX d 1-5; MTX weekly d 8-78; MP d 1-84; IT MTX d 1 Arm D: VIN d 1; DEX d 1-5; HD MTX weekly d 8-78; MP d 1-84; IT MTX d 1
Arm/Group | B-ALL Average Risk: MTX 20 mg/m^2/Week Starting Dose | B-ALL Average Risk: MTX 40 mg/m^2/Week Starting Dose
Number analyzed (Participants) | 1186 | 1178
percent probability | 95.05 [93.27 to 96.83] | 94.17 [92.23 to 96.11]

2. Primary Outcome: DFS in Average Risk (AR) Patients Based on the Pulse Frequency Randomization
Description: as for outcome 1
Time Frame: 5.7 years
Population: Average Risk (AR) B-ALL patients who were randomized and started maintenance
Measure: Number (95% Confidence Interval); unit: percent probability
Groups:
- B-ALL Average Risk: VCR/DEX Pulse Every 4 Weeks; B-ALL Average Risk: VCR/DEX Pulse Every 12 Weeks: Cons. (4 wks): vincristine (VIN) day (d) 1; mercaptopurine (MP) d 1-28; IT MTX d 1/8/15; leucovorin (LV) d 3-4/10-11/17-18 Int. maint. I (8 wks): VIN and MTX d 1/11/21/31/41; IT MTX d 31; LV d 33-34 Delayed-intensification (8 wks): dexamethasone (DEX) d 1-7/15-21; VIN and doxorubicin d 1/8/15; pegaspargase d 4; cyclophosphamide d 29; thioguanine d 29-42; cytarabine d 29-32/33-39; IT MTX d 1/29; LV d 3-4/31-32 Int. maint. II (8 wks): VIN and MTX d 1/11/21/31/41; IT MTX d 1/31; LV d 3-4/33-34 Maintenance: repeat every 12 wks for 2 yrs (girls), 3 yrs (boys) from start IM1 Arm A: VIN d 1/29/57; DEX d 1-5/29-33/57-61; MTX weekly d 8-78; MP d 1-84; and IT MTX d 1 Arm B: VIN d 1/29/57; DEX d 1-5/29-33/57-61; high-dose (HD) MTX weekly d 8-78; MP d 1-84; and IT MTX d 1 Arm C: VIN d 1; DEX d 1-5; MTX weekly d 8-78; MP d 1-84; IT MTX d 1 Arm D: VIN d 1; DEX d 1-5; HD MTX weekly d 8-78; MP d 1-84; IT MTX d 1
Arm/Group | B-ALL Average Risk: VCR/DEX Pulse Every 4 Weeks | B-ALL Average Risk: VCR/DEX Pulse Every 12 Weeks
Number analyzed (Participants) | 1186 | 1178
percent probability | 94.10 [92.16 to 96.04] | 95.13 [93.35 to 96.91]

3. Primary Outcome: DFS in Low Risk (LR) Patients Based on Randomization to 1 of 2 Low-intensity Regimens
Description: DFS is calculated as the time from randomization at the end of Induction to first event (relapse, second malignancy, remission death) or date of last contact. Five year DFS estimates will be calculated from the point of randomization for both groups. Two-sided 95% confidence intervals will be calculated.
Time Frame: 5.1 years
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | B-ALL Low Risk Arm I (LR-M) | B-ALL Low Risk Arm II (LR-C)
Number analyzed (Participants) | 301 | 302
percent probability | 98.75 [97.14 to 100.00] | 98.50 [96.75 to 100.00]

4. Primary Outcome: DFS for SR Down Syndrome Patients With Standardized Treatment and Enhanced Supportive Care
Description: DFS is calculated as the time from end of Induction to first event (relapse, second malignancy, remission death) or date of last contact. The 5-year DFS and 95% confidence interval for these patients will be estimated.
Time Frame: 5.1 years
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Standard Risk With Down Syndrome
Number analyzed (Participants) | 224
percent probability | 89.77 [83.60 to 95.94]

5. Primary Outcome: Sample Collection of Central Path Review Slides in B-LLy Patients
Description: Percent of B-LLy patients who had adequate/usable samples of samples collected will be reported.
Time Frame: Up to 1 month
Population: patients who had samples collected near diagnosis
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | B-LLy
Number analyzed (Participants) | 39
percentage of patients | 89.7 [80.2 to 99.3]

6. Primary Outcome: Event Free Survival (EFS) for B-LLy Patients
Description: EFS is calculated as the Time from study enrollment to first event (induction failure, relapse, second malignancy, remission death) or date of last contact. The 5-year EFS and 95% confidence interval for these patients will be estimated.
Time Frame: 5 years
Population: Ineligible patients are excluded
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | B-LLy
Number analyzed (Participants) | 48
percent probability | 94.54 [78.17 to 100.00]

7. Primary Outcome: Overall Survival (OS) for B-LLy Patients
Description: OS is calculated as the time from study enrollment to death or date of last contact. The 5-year OS and 95% confidence interval for these patients will be estimated.
Time Frame: 5 years
Population: Ineligible patients are excluded
Measure: Number (95% Confidence Interval); unit: percent probability
Groups:
- B-LLy: Induction: same trt as B-ALL Consolidation (4 wks): vincristine sulfate day 1; mercaptopurine days 1-28; IT methotrexate (MTX) days 1/8/15; leucovorin calcium days 3-4,10-11,17-18 Interim maintenance I (8 wks): vincristine sulfate and MTX 2-15 min days 1/11/21/31/41; IT MTX day 31; leucovorin calcium days 33-34 Delayed-intensification (8 wks): dexamethasone days 1-7 and 15-21; vincristine sulfate and doxorubicin hydrochloride on days 1/8/15; pegaspargase 1-2 hrs day 4; cyclophosphamide day 29; thioguanine days 29-42; cytarabine 29-32, 33-39; IT MTX days 1/29; and leucovorin calcium days 3-4, 31-32 Interim maintenance II (8 wks): vincristine sulfate and MTX days 1/11/21/31/41; IT MTX days 1/31; and leucovorin calcium days 3-4, 33/34 Maintenance: vincristine sulfate day 1; dexamethasone days 1-5; MTX weekly days 8-78; mercaptopurine days 1-84; and IT MTX day 1. Courses repeat every 4 wks for 2 yrs (from the start of IMI therapy).
Arm/Group | B-LLy
Number analyzed (Participants) | 48
percent probability | 93.97 [76.88 to 100.00]

8. Secondary Outcome: Burden of Therapy in AR Patients Overall at End of Consolidation Therapy: Emotional
Description: Age standardized Quality of life, measured by the emotional subscale of Pediatric Quality of Life Inventory 4.0 Generic Core Scales (PedsQL), will be calculated with mean and standard deviation reported.
Time Frame: 2 Months
Population: AR patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Groups:
- B-ALL Average Risk: Cons. (4 wks): vincristine (VIN) day (d) 1; mercaptopurine (MP) d 1-28; IT MTX d 1/8/15; leucovorin (LV) d 3-4/10-11/17-18 Int. maint. I (8 wks): VIN and MTX d 1/11/21/31/41; IT MTX d 31; LV d 33-34 Delayed-intensification (8 wks): dexamethasone (DEX) d 1-7/15-21; VIN and doxorubicin d 1/8/15; pegaspargase d 4; cyclophosphamide d 29; thioguanine d 29-42; cytarabine d 29-32/33-39; IT MTX d 1/29; LV d 3-4/31-32 Int. maint. II (8 wks): VIN and MTX d 1/11/21/31/41; IT MTX d 1/31; LV d 3-4/33-34 Maintenance: repeat every 12 wks for 2 yrs (girls), 3 yrs (boys) from start IM1 Arm A: VIN d 1/29/57; DEX d 1-5/29-33/57-61; MTX weekly d 8-78; MP d 1-84; and IT MTX d 1 Arm B: VIN d 1/29/57; DEX d 1-5/29-33/57-61; high-dose (HD) MTX weekly d 8-78; MP d 1-84; and IT MTX d 1 Arm C: VIN d 1; DEX d 1-5; MTX weekly d 8-78; MP d 1-84; IT MTX d 1 Arm D: VIN d 1; DEX d 1-5; HD MTX weekly d 8-78; MP d 1-84; IT MTX d 1
Arm/Group | B-ALL Average Risk
Number analyzed (Participants) | 379
Z-Score | -1.21 (1.14)

9. Secondary Outcome: Burden of Therapy in AR Patients Overall at End of Maintenance Cycle 1: Emotional
Description: as for outcome 8
Time Frame: 1 year
Population: AR patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk
Number analyzed (Participants) | 242
Z-Score | -0.86 (1.10)

10. Secondary Outcome: Burden of Therapy in AR Patients Overall at End of Maintenance Cycle 4: Emotional
Description: as for outcome 8
Time Frame: 1.7 years
Population: AR patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk
Number analyzed (Participants) | 221
Z-Score | -0.84 (1.11)

11. Secondary Outcome: Burden of Therapy in AR Patients Overall at End of Maintenance Cycle 7 (Boys)/End of Therapy (Girls): Emotional
Description: as for outcome 8
Time Frame: 2.5 years
Population: AR patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk
Number analyzed (Participants) | 209
Z-Score | -0.74 (1.10)

12. Secondary Outcome: Burden of Therapy in Boy AR Patients Overall at End of Therapy: Emotional
Description: Age standardized Quality of life, measured by the emotional subscale of Pediatric Quality of Life Inventory 4.0 Genetic Core Scales (PedsQL), will be calculated with mean and standard deviation reported.
Time Frame: 3.2 years
Population: AR boy patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk
Number analyzed (Participants) | 80
Z-Score | -0.62 (1.26)

13. Secondary Outcome: Burden of Therapy in AR Patients Overall at End of Consolidation Therapy: Physical
Description: Age and gender standardized Quality of life, measured by the physical subscale of Pediatric Quality of Life Inventory 4.0 Generic Core Scales (PedsQL), will be calculated with mean and standard deviation reported.
Time Frame: 2 Months
Population: AR patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk
Number analyzed (Participants) | 379
Z-Score | -1.44 (1.10)

14. Secondary Outcome: Burden of Therapy in AR Patients Overall at End of Maintenance Cycle 1: Physical
Description: Age standardized Quality of life, measured by the physical subscale of Pediatric Quality of Life Inventory 4.0 Generic Core Scales (PedsQL), will be calculated with mean and standard deviation reported.
Time Frame: 1 Year
Population: AR patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk
Number analyzed (Participants) | 242
Z-Score | -0.59 (1.02)

15. Secondary Outcome: Burden of Therapy in AR Patients Overall at End of Maintenance Cycle 4: Physical
Description: as for outcome 14
Time Frame: 1.7 years
Population: AR patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk
Number analyzed (Participants) | 221
Z-Score | -0.63 (1.06)

16. Secondary Outcome: Burden of Therapy in AR Patients Overall at End of Maintenance Cycle 7 (Boys)/End of Therapy (Girls): Physical
Description: as for outcome 14
Time Frame: 2.4 Years
Population: AR patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk
Number analyzed (Participants) | 209
Z-Score | -0.66 (1.15)

17. Secondary Outcome: Burden of Therapy in Boy AR Patients Overall at End of Therapy: Physical
Description: as for outcome 14
Time Frame: 3.2 years
Population: AR boy patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk
Number analyzed (Participants) | 80
Z-Score | -0.67 (1.23)

18. Secondary Outcome: Burden of Therapy in AR Patients Overall at End of Consolidation Therapy: School
Description: Age standardized Quality of life, measured by the school subscale of Pediatric Quality of Life Inventory 4.0 Generic Core Scales (PedsQL), will be calculated with mean and standard deviation reported.
Time Frame: 2 Months
Population: Data are unavailable
Arm/Group | B-ALL Average Risk
Number analyzed (Participants) | 0

19. Secondary Outcome: Burden of Therapy in AR Patients Overall at End of Maintenance Cycle 1: School
Description: as for outcome 18
Time Frame: 1 Year
Population: Data are unavailable
Arm/Group | B-ALL Average Risk
Number analyzed (Participants) | 0

20. Secondary Outcome: Burden of Therapy in AR Patients Overall at End of Maintenance Cycle 4: School
Description: as for outcome 18
Time Frame: 1.7 Years
Population: Data are unavailable
Arm/Group | B-ALL Average Risk
Number analyzed (Participants) | 0

21. Secondary Outcome: Burden of Therapy in AR Patients Overall at End of Maintenance Cycle 7 (Boys)/End of Therapy (Girls): School
Description: as for outcome 18
Time Frame: 2.4 years
Population: Data are unavailable
Arm/Group | B-ALL Average Risk
Number analyzed (Participants) | 0

22. Secondary Outcome: Burden of Therapy in Boy AR Patients Overall at End of Therapy: School
Description: as for outcome 18
Time Frame: 3.2 Years
Population: Data are unavailable
Arm/Group | B-ALL Average Risk
Number analyzed (Participants) | 0

23. Secondary Outcome: Burden of Therapy in AR Patients Overall at End of Consolidation Therapy: Social Functioning
Description: Age standardized Quality of life, measured by the social functioning subscale of Pediatric Quality of Life Inventory 4.0 Generic Core Scales (PedsQL), will be calculated with mean and standard deviation reported.
Time Frame: 2 Months
Population: AR patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk
Number analyzed (Participants) | 379
Z-Score | -0.42 (0.84)

24. Secondary Outcome: Burden of Therapy in AR Patients Overall at End of Maintenance Cycle 1: Social Functioning
Description: as for outcome 23
Time Frame: 1 Year
Population: AR patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk
Number analyzed (Participants) | 242
Z-Score | -0.19 (0.92)

25. Secondary Outcome: Burden of Therapy in AR Patients Overall at End of Maintenance Cycle 4: Social Functioning
Description: as for outcome 23
Time Frame: 1.7 Years
Population: AR patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk
Number analyzed (Participants) | 221
Z-Score | -0.20 (0.94)

26. Secondary Outcome: Burden of Therapy in AR Patients Overall at End of Maintenance Cycle 7 (Boys)/End of Therapy (Girls): Social Functioning
Description: as for outcome 23
Time Frame: 2.4 Years
Population: AR patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk
Number analyzed (Participants) | 209
Z-Score | -0.30 (0.97)

27. Secondary Outcome: Burden of Therapy in Boy AR Patients Overall at End of Therapy: Social Functioning
Description: as for outcome 23
Time Frame: 3.2 Years
Population: AR boy patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk
Number analyzed (Participants) | 80
Z-Score | -0.40 (1.17)

28. Secondary Outcome: Burden of Therapy in AR Patients by Vincristine Pulse Frequency Randomization Groups (4 Week vs. 12 Week) at End of Maintenance Cycle 4: Emotional
Description: Age standardized Quality of life, measured by the emotional subscale of Pediatric Quality of Life Inventory 4.0 Generic Core Scales (PedsQL), will be calculated for each group with means and standard deviation reported.
Time Frame: 1.7 years
Population: AR patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk: VCR/DEX Pulse Every 4 Weeks | B-ALL Average Risk: VCR/DEX Pulse Every 12 Weeks
Number analyzed (Participants) | 122 | 99
Z-Score | -0.80 (1.11) | -0.89 (1.13)

29. Secondary Outcome: Burden of Therapy in AR Patients by Vincristine Pulse Frequency Randomization Groups (4 Week vs. 12 Week) at End of Maintenance Cycle 7 (Boys)/End of Therapy (Girls): Emotional
Description: Age standardized Quality of life, measured by the emotional subscale of Pediatric Quality of Life Inventory 4.0 Generic Core Scales (PedsQL), will be calculated for each group with mean and standard deviation reported.
Time Frame: 2.4 Years
Population: AR patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk: VCR/DEX Pulse Every 4 Weeks | B-ALL Average Risk: VCR/DEX Pulse Every 12 Weeks
Number analyzed (Participants) | 111 | 98
Z-Score | -0.72 (1.10) | -0.77 (1.11)

30. Secondary Outcome: Burden of Therapy in Boy AR Patients by Vincristine Pulse Frequency Randomization Groups (4 Week vs. 12 Week) at End of Therapy: Emotional
Description: as for outcome 29
Time Frame: 3.2 Years
Population: AR boy patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk: VCR/DEX Pulse Every 4 Weeks | B-ALL Average Risk: VCR/DEX Pulse Every 12 Weeks
Number analyzed (Participants) | 43 | 37
Z-Score | -0.71 (1.45) | -0.51 (1.00)

31. Secondary Outcome: Burden of Therapy in AR Patients by Vincristine Pulse Frequency Randomization Groups (4 Week vs. 12 Week) at End of Maintenance Cycle 4: Physical
Description: Age standardized Quality of life, measured by the physical subscale of Pediatric Quality of Life Inventory 4.0 Generic Core Scales (PedsQL), will be calculated for each group with means and standard deviation reported.
Time Frame: 1.7 Years
Population: AR patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk: VCR/DEX Pulse Every 4 Weeks | B-ALL Average Risk: VCR/DEX Pulse Every 12 Weeks
Number analyzed (Participants) | 122 | 99
Z-Score | -0.62 (1.01) | -0.64 (1.11)

32. Secondary Outcome: Burden of Therapy in AR Patients by Vincristine Pulse Frequency Randomization Groups (4 Week vs. 12 Week) at End of Maintenance Cycle 7 (Boys)/End of Therapy (Girls): Physical
Description: Age standardized Quality of life, measured by the physical subscale of Pediatric Quality of Life Inventory 4.0 Generic Core Scales (PedsQL), will be calculated for each group with mean and standard deviation reported.
Time Frame: 2.4 Years
Population: AR patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk: VCR/DEX Pulse Every 4 Weeks | B-ALL Average Risk: VCR/DEX Pulse Every 12 Weeks
Number analyzed (Participants) | 111 | 98
Z-Score | -0.64 (1.11) | -0.67 (1.19)

33. Secondary Outcome: Burden of Therapy in Boy AR Patients by Vincristine Pulse Frequency Randomization Groups (4 Week vs. 12 Week) at End of Therapy: Physical
Description: as for outcome 32
Time Frame: 3.2 Years
Population: AR boy patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk: VCR/DEX Pulse Every 4 Weeks | B-ALL Average Risk: VCR/DEX Pulse Every 12 Weeks
Number analyzed (Participants) | 43 | 37
Z-Score | -0.85 (1.30) | -0.47 (1.13)

34. Secondary Outcome: Burden of Therapy in AR Patients by Vincristine Pulse Frequency Randomization Groups (4 Week vs. 12 Week) at End of Maintenance Cycle 4: School
Description: Age standardized Quality of life, measured by the school subscale of Pediatric Quality of Life Inventory 4.0 Generic Core Scales (PedsQL), will be calculated for each group with means and standard deviation reported.
Time Frame: 1.7 Years
Population: Data are unavailable
Arm/Group | B-ALL Average Risk: VCR/DEX Pulse Every 4 Weeks | B-ALL Average Risk: VCR/DEX Pulse Every 12 Weeks
Number analyzed (Participants) | 0 | 0

35. Secondary Outcome: Burden of Therapy in AR Patients by Vincristine Pulse Frequency Randomization Groups (4 Week vs. 12 Week) at End of Maintenance Cycle 7 (Boys)/End of Therapy (Girls): School
Description: Age standardized Quality of life, measured by the school subscale of Pediatric Quality of Life Inventory 4.0 Generic Core Scales (PedsQL), will be calculated for each group with mean and standard deviation reported.
Time Frame: 2.4 Years
Population: Data are unavailable
Arm/Group | B-ALL Average Risk: VCR/DEX Pulse Every 4 Weeks | B-ALL Average Risk: VCR/DEX Pulse Every 12 Weeks
Number analyzed (Participants) | 0 | 0

36. Secondary Outcome: Burden of Therapy in Boy AR Patients by Vincristine Pulse Frequency Randomization Groups (4 Week vs. 12 Week) at End of Therapy: School
Description: as for outcome 35
Time Frame: 3.2 Years
Population: Data are unavailable
Arm/Group | B-ALL Average Risk: VCR/DEX Pulse Every 4 Weeks | B-ALL Average Risk: VCR/DEX Pulse Every 12 Weeks
Number analyzed (Participants) | 0 | 0

37. Secondary Outcome: Burden of Therapy in AR Patients by Vincristine Pulse Frequency Randomization Groups (4 Week vs. 12 Week) at End of Maintenance Cycle 4: Social Functioning
Description: Age standardized Quality of life, measured by the social functioning subscale of Pediatric Quality of Life Inventory 4.0 Generic Core Scales (PedsQL), will be calculated for each group with means and standard deviation reported.
Time Frame: 1.7 Years
Population: AR patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk: VCR/DEX Pulse Every 4 Weeks | B-ALL Average Risk: VCR/DEX Pulse Every 12 Weeks
Number analyzed (Participants) | 122 | 99
Z-Score | -0.16 (0.85) | -0.25 (1.03)

38. Secondary Outcome: Burden of Therapy in AR Patients by Vincristine Pulse Frequency Randomization Groups (4 Week vs. 12 Week) at End of Maintenance Cycle 7 (Boys)/End of Therapy (Girls): Social Functioning
Description: Age standardized Quality of life, measured by the social functioning subscale of Pediatric Quality of Life Inventory 4.0 Generic Core Scales (PedsQL), will be calculated for each group with mean and standard deviation reported.
Time Frame: 2.4 Years
Population: AR patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk: VCR/DEX Pulse Every 4 Weeks | B-ALL Average Risk: VCR/DEX Pulse Every 12 Weeks
Number analyzed (Participants) | 111 | 98
Z-Score | -0.27 (0.95) | -0.34 (1.00)

39. Secondary Outcome: Burden of Therapy in Boy AR Patients by Vincristine Pulse Frequency Randomization Groups (4 Week vs. 12 Week) at End of Therapy: Social Functioning
Description: as for outcome 38
Time Frame: 3.2 Years
Population: AR boy patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk: VCR/DEX Pulse Every 4 Weeks | B-ALL Average Risk: VCR/DEX Pulse Every 12 Weeks
Number analyzed (Participants) | 43 | 37
Z-Score | -0.46 (1.20) | -0.33 (1.15)

40. Secondary Outcome: Characterize Vincristine-associated Neuropathy in Children Undergoing Therapy for Average Risk (AR) ALL at End of Consolidation Therapy-Right
Description: Strength in the right ankle dorsiflexors averaged over two measurements. Age and gender standardized mean and standard deviation for the cohort will be reported.
Time Frame: 2 Months
Population: AR patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk
Number analyzed (Participants) | 90
Z-Score | -0.87 (1.67)

41. Secondary Outcome: Characterize Vincristine-associated Neuropathy in Children Undergoing Therapy for Average Risk (AR) ALL at End of Consolidation Therapy-Left
Description: Strength in the left ankle dorsiflexors averaged over two measurements. Age and gender standardized mean and standard deviation for the cohort will be reported.
Time Frame: 2 Months
Population: AR patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk
Number analyzed (Participants) | 89
Z-Score | -0.84 (1.85)

42. Secondary Outcome: Characterize Vincristine-associated Neuropathy in Children Undergoing Therapy for Average Risk (AR) ALL at End of Maintenance Cycle 1: Right
Description: as for outcome 40
Time Frame: 1 Year
Population: AR patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk
Number analyzed (Participants) | 89
Z-Score | -0.39 (2.10)

43. Secondary Outcome: Characterize Vincristine-associated Neuropathy in Children Undergoing Therapy for Average Risk (AR) ALL at End of Maintenance Cycle 1: Left
Description: as for outcome 41
Time Frame: 1 Year
Population: AR patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk
Number analyzed (Participants) | 88
Z-Score | -0.36 (1.97)

44. Secondary Outcome: Characterize Vincristine-associated Neuropathy in Children Undergoing Therapy for Average Risk (AR) ALL at End of Maintenance Cycle 7 (Boys)/End of Therapy (Girls): Right
Description: as for outcome 40
Time Frame: 2.4 Years
Population: AR patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk
Number analyzed (Participants) | 59
Z-Score | -0.27 (2.06)

45. Secondary Outcome: Characterize Vincristine-associated Neuropathy in Children Undergoing Therapy for Average Risk (AR) ALL at End of Maintenance Cycle 7 (Boys)/End of Therapy (Girls): Left
Description: as for outcome 41
Time Frame: 2.4 Years
Population: AR patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk
Number analyzed (Participants) | 58
Z-Score | -0.28 (2.00)

46. Secondary Outcome: Characterize Vincristine-associated Neuropathy in Children Undergoing Therapy for Average Risk (AR) ALL 12 Months Post Therapy: Right
Description: as for outcome 40
Time Frame: 4.2 Years
Population: AR patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk
Number analyzed (Participants) | 35
Z-Score | -1.12 (2.27)

47. Secondary Outcome: Characterize Vincristine-associated Neuropathy in Children Undergoing Therapy for Average Risk (AR) ALL 12 Months Post Therapy: Left
Description: as for outcome 41
Time Frame: 4.2 Years
Population: AR patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk
Number analyzed (Participants) | 35
Z-Score | -1.19 (2.14)

48. Secondary Outcome: Characterize Vincristine-associated Neuropathy in Children Undergoing Therapy for Average Risk (AR) ALL by Vincristine Pulse Frequency Randomization Groups (4 Week vs. 12 Week) at End of Maintenance Cycle 7 (Boys)/End of Therapy (Girls): Right
Description: Strength in the right ankle dorsiflexors averaged over two measurements. Age and gender standardized mean and standard deviation for each randomization group will be reported.
Time Frame: 2.4 Years
Population: AR patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Groups:
- B-ALL Average Risk: VCR/DEX Pulse Every 4 Weeks; B-ALL Average Risk: VCR/DEX Pulse Every 12 Weeks: Cons. (4 wks): vincristine (VIN) day (d) 1; mercaptopurine (MP) d 1-28; IT MTX d 1/8/15; leucovorin (LV) d 3-4/10-11/17-18 Int. maint. I (8 wks): VIN and MTX d 1/11/21/31/41; IT MTX d 31; LV d 33-34 Delayedintensification (8 wks): dexamethasone (DEX) d 1-7/15-21; VIN and doxorubicin d 1/8/15; pegaspargase d 4; cyclophosphamide d 29; thioguanine d 29-42; cytarabine d 29-32/33-39; IT MTX d 1/29; LV d 3-4/31-32 Int.
  maint. II (8 wks): VIN and MTX d 1/11/21/31/41; IT MTX d 1/31; LV d 3-4/33-34 Maintenance: repeat every 12 wks for 2 yrs (girls), 3 yrs (boys) from start IM1 Arm A: VIN d 1/29/57; DEX d 1-5/29-33/57-61; MTX weekly d 8-78; MP d 1-84; and IT MTX d 1 Arm B: VIN d 1/29/57; DEX d 1-5/29-33/57-61; high-dose (HD) MTX weekly d 8-78; MP d 1-84; and IT MTX d 1 Arm C: VIN d 1; DEX d 1-5; MTX weekly d 8-78; MP d 1-84; IT MTX d 1 Arm D: VIN d 1; DEX d 1-5; HD MTX weekly d 8-78; MP d 1-84; IT MTX d 1
Arm/Group | B-ALL Average Risk: VCR/DEX Pulse Every 4 Weeks | B-ALL Average Risk: VCR/DEX Pulse Every 12 Weeks
Number analyzed (Participants) | 35 | 40
Z-Score | -1.12 (2.27) | -0.02 (3.01)

49. Secondary Outcome: Characterize Vincristine-associated Neuropathy in Children Undergoing Therapy for Average Risk (AR) ALL by Vincristine Pulse Frequency Randomization Groups (4 Week vs. 12 Week) at End of Maintenance Cycle 7 (Boys)/End of Therapy (Girls): Left
Description: Strength in the left ankle dorsiflexors averaged over two measurements. Age and gender standardized mean and standard deviation for each randomization group will be reported.
Time Frame: 2.4 Years
Population: AR patients who had data collected
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | B-ALL Average Risk: VCR/DEX Pulse Every 4 Weeks | B-ALL Average Risk: VCR/DEX Pulse Every 12 Weeks
Number analyzed (Participants) | 35 | 40
Z-Score | -1.19 (2.14) | 0.21 (2.99)

ADVERSE EVENTS:
Time Frame: Up to 9 years
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution, via expedited reporting (NCI AdEERs / CAeRs). The "AE Other" table reflects all CTCAEs collected excluding those that were reported as SAEs. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | B-ALL | B-LLy | B-ALL Average Risk | Standard Risk With Down Syndrome | B-ALL Low Risk Arm I (LR-M) | B-ALL Low Risk Arm II (LR-C) | B-ALL Average Risk-Arm A | B-ALL Average Risk-Arm B | B-ALL Average Risk-Arm C | B-ALL Average Risk-Arm D
All-Cause Mortality (participants affected / at risk) | 125/9229 | 2/48 | 16/3122 | 11/224 | 0/301 | 1/302 | 7/600 | 8/586 | 6/586 | 7/592
Serious Adverse Events (participants affected / at risk) | 72/9229 | 0/48 | 16/3122 | 9/224 | 0/301 | 0/302 | 7/600 | 7/586 | 4/586 | 3/592
Other Adverse Events (participants affected / at risk) | 1776/9229 | 30/48 | 1037/3122 | 191/224 | 103/301 | 143/302 | 180/600 | 204/586 | 156/586 | 152/592
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | B-ALL (N=9229) | B-LLy (N=48) | B-ALL Average Risk (N=3122) | Standard Risk With Down Syndrome (N=224) | B-ALL Low Risk Arm I (LR-M) (N=301) | B-ALL Low Risk Arm II (LR-C) (N=302) | B-ALL Average Risk-Arm A (N=600) | B-ALL Average Risk-Arm B (N=586) | B-ALL Average Risk-Arm C (N=586) | B-ALL Average Risk-Arm D (N=592)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic necrosis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death NOS (General disorders) | 7 (7) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Multi-organ failure (General disorders) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sudden death NOS (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Anaphylaxis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune system disorders - Other, specify (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cecal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 4 (4) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 5 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periorbital infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritoneal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 23 (23) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cholesterol high (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema cerebral (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Personality change (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | B-ALL (N=9229) | B-LLy (N=48) | B-ALL Average Risk (N=3122) | Standard Risk With Down Syndrome (N=224) | B-ALL Low Risk Arm I (LR-M) (N=301) | B-ALL Low Risk Arm II (LR-C) (N=302) | B-ALL Average Risk-Arm A (N=600) | B-ALL Average Risk-Arm B (N=586) | B-ALL Average Risk-Arm C (N=586) | B-ALL Average Risk-Arm D (N=592)
Anemia (Blood and lymphatic system disorders) | 26 (26) | 0 (0) | 19 (21) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 2 (2) | 2 (2) | 3 (3)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 114 (114) | 0 (0) | 101 (112) | 114 (185) | 13 (15) | 14 (16) | 28 (34) | 35 (40) | 23 (26) | 27 (32)
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wolff-Parkinson-White syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Congenital, familial and genetic disorders - Other, specify (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cushingoid (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocrine disorders - Other, specify (Endocrine disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Optic nerve disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous hemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 8 (8) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Anal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Cecal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 6 (6) | 0 (0) | 7 (8) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 13 (13) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 8 (8) | 0 (0) | 12 (12) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric necrosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileal perforation (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 34 (34) | 0 (0) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Jejunal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jejunal perforation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 70 (70) | 16 (17) | 354 (374) | 88 (120) | 21 (25) | 38 (46) | 18 (19) | 22 (25) | 15 (16) | 12 (13)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 90 (90) | 0 (0) | 15 (15) | 1 (1) | 0 (0) | 4 (8) | 5 (8) | 2 (2) | 3 (8) | 4 (5)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 15 (15) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 8 (9) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 18 (18) | 0 (0) | 36 (43) | 4 (4) | 6 (6) | 2 (2) | 7 (10) | 3 (4) | 6 (6) | 8 (10)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Localized edema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 8 (8) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gallbladder pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 0 (0) | 7 (7) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 22 (22) | 1 (1) | 50 (50) | 1 (1) | 0 (0) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylaxis (Immune system disorders) | 9 (9) | 2 (2) | 21 (21) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Immune system disorders - Other, specify (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorectal infection (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Appendicitis perforated (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (3) | 9 (9) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Catheter related infection (Infections and infestations) | 44 (44) | 0 (0) | 6 (6) | 8 (11) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Cecal infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 5 (5) | 0 (0) | 1 (1) | 4 (6) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Encephalitis infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocarditis infective (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 7 (7) | 0 (0) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Esophageal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gum infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 122 (125) | 2 (2) | 48 (50) | 62 (77) | 6 (6) | 5 (6) | 12 (12) | 6 (7) | 13 (14) | 11 (12)
Infective myositis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 19 (19) | 1 (1) | 13 (13) | 42 (53) | 5 (5) | 0 (0) | 6 (6) | 6 (6) | 2 (2) | 3 (3)
Lymph gland infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mediastinal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 5 (5) | 0 (0) | 3 (3) | 9 (9) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 3 (3) | 0 (0) | 6 (6) | 9 (9) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 6 (7)
Pancreas infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papulopustular rash (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Periorbital infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral nerve infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritoneal infection (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scrotal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 100 (100) | 2 (2) | 22 (22) | 5 (5) | 2 (3) | 2 (2) | 6 (6) | 10 (10) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 4 (4) | 1 (2) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 19 (19) | 0 (0) | 3 (4) | 22 (25) | 1 (1) | 1 (1) | 2 (2) | 4 (5) | 2 (2) | 2 (2)
Small intestine infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 12 (12) | 0 (0) | 23 (24) | 49 (66) | 4 (8) | 5 (5) | 7 (8) | 8 (10) | 6 (6) | 10 (13)
Urethral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 8 (8) | 0 (0) | 10 (11) | 11 (15) | 2 (3) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 4 (4)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 14 (14) | 0 (0) | 0 (0) | 5 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheal obstruction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 16 (16) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 195 (195) | 6 (7) | 139 (160) | 22 (31) | 29 (45) | 28 (38) | 42 (56) | 46 (61) | 36 (43) | 37 (51)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 8 (8) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 72 (73) | 3 (3) | 22 (23) | 9 (9) | 5 (5) | 5 (6) | 11 (12) | 5 (5) | 7 (8) | 6 (7)
Blood bilirubin increased (Investigations) | 111 (111) | 9 (10) | 9 (9) | 12 (16) | 20 (25) | 16 (18) | 37 (40) | 36 (49) | 33 (61) | 32 (44)
Cholesterol high (Investigations) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibrinogen decreased (Investigations) | 55 (55) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GGT increased (Investigations) | 34 (34) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Investigations - Other, specify (Investigations) | 3 (3) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 39 (40) | 0 (0) | 10 (10) | 2 (2) | 1 (1) | 2 (2) | 2 (3) | 2 (2) | 2 (2) | 4 (5)
Lymphocyte count decreased (Investigations) | 13 (13) | 0 (0) | 6 (6) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 333 (339) | 1 (1) | 201 (259) | 102 (203) | 14 (25) | 23 (31) | 27 (43) | 40 (59) | 29 (38) | 39 (58)
Platelet count decreased (Investigations) | 161 (161) | 1 (1) | 38 (40) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 2 (3) | 0 (0) | 3 (3)
Serum amylase increased (Investigations) | 13 (14) | 0 (0) | 6 (6) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Weight gain (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 141 (142) | 0 (0) | 41 (44) | 4 (5) | 3 (3) | 4 (4) | 1 (1) | 6 (7) | 3 (3) | 5 (6)
Acidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 4 (4) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 6 (6) | 1 (1) | 13 (13) | 7 (7) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 2 (3)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 147 (147) | 0 (0) | 5 (6) | 4 (5) | 3 (3) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 10 (10) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 24 (24) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 8 (8) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 (8) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 41 (41) | 0 (0) | 7 (7) | 4 (4) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 4 (4) | 4 (4) | 6 (7) | 4 (4) | 6 (6)
Hypokalemia (Metabolism and nutrition disorders) | 79 (79) | 1 (1) | 34 (40) | 8 (8) | 3 (3) | 7 (7) | 4 (5) | 7 (7) | 3 (4) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 22 (22) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 10 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1) | 5 (5) | 3 (3) | 3 (3) | 6 (6) | 6 (6) | 10 (10) | 7 (8) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue necrosis lower limb (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue necrosis upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Akathisia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arachnoiditis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Central nervous system necrosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 13 (13) | 1 (1) | 7 (7) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 5 (6) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 17 (17) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukoencephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Movements involuntary (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 5 (6) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oculomotor nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 175 (175) | 2 (2) | 98 (109) | 14 (15) | 4 (4) | 9 (9) | 8 (13) | 14 (17) | 5 (5) | 4 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 151 (151) | 3 (4) | 69 (83) | 7 (7) | 5 (8) | 9 (15) | 10 (20) | 17 (27) | 8 (8) | 7 (7)
Recurrent laryngeal nerve palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 10 (10) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 69 (69) | 4 (4) | 52 (59) | 2 (2) | 3 (3) | 4 (4) | 6 (12) | 3 (3) | 4 (4) | 10 (11)
Stroke (Nervous system disorders) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Personality change (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychosis (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 16 (16) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal calculi (Renal and urinary disorders) | 13 (13) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scrotal pain (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial stricture (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 0 (0) | 3 (3) | 9 (10) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 19 (19) | 0 (0) | 4 (4) | 6 (6) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 3 (3)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 26 (26) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 18 (18) | 0 (0) | 6 (6) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Peripheral ischemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 55 (56) | 2 (2) | 15 (17) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular disorders - Other, specify (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/30/NCT01190930/Prot_SAP_000.pdf